CLINICAL TRIAL: NCT07403604
Title: Human Models of Selective Insulin Resistance: Diazoxide, Part I
Brief Title: Effect of Insulin Lowering on Lipogenesis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: University of California, Berkeley (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Joshua Cook, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: AAAV7588; K23DK140614 (NIH)
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Hyperinsulinemia; Insulin Resistance; Non-Alcoholic Fatty Liver Disease; Prediabetic State; Obesity
Keywords: Hyperinsulinemia; Insulin Resistance; Metabolic Dysfunction-Associated Steatotic Liver Disease; Non-Alcoholic Fatty Liver Disease; Triglycerides
MeSH Terms: conditions — Hyperinsulinism; Insulin Resistance; Non-alcoholic Fatty Liver Disease; Prediabetic State; Obesity | interventions — Diazoxide; Deuterium Oxide

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of two study groups. All participants will receive a 1-week placebo treatment, while 4-12 weeks later, one group will receive diazoxide for 1 week while the other will receive a second week of placebo.
Who Masked: Participant, Investigator
Masking Description: Participants will be masked to treatment during both 1-week study periods, while investigators will be masked only during the second 1-week study period, when participants will receive either diazoxide or placebo. Routine unblinding will occur to investigators only after all of a participant's samples have been submitted for laboratory analysis. It should be noted that investigators may get a sense of group allocation based on changes in blood glucose. However, due to interindividual variability in extent of insulin resistance and body mass index, it will not be possible to assuredly decode the randomization prior to unblinding. The blinding of the study Principal Investigator (PI) will be repealed only in the case of early withdrawal and/or medical emergency (e.g., severe hyperglycemia), which in most cases will result in study termination anyway. Participants will be notified of their group assignment once all relevant data are collected and analyzed if opted in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Placebo first, then Diazoxide (Experimental): During the first 1-week study period, participants will ingest a placebo solution at 14 doses over 7 days. During the second 1-week study period, 4-12 weeks later, participants will ingest diazoxide oral suspension at 2 mg per kg body weight per dose (14 doses over 7 days). Blinding will occur by completely covering single-dose oral syringes with labels. 80% of participants will be randomized to this arm.
  Interventions: Drug: Placebo; Drug: Diazoxide Oral Suspension, 2 mg per kg per dose; Drug: Deuterated water (2H2O/D2O), 70%; Diagnostic Test: Insulin Suppression Test (IST)
- Placebo / Placebo (Placebo Comparator): During the first 1-week study period, participants will ingest a placebo solution at 14 doses over 7 days. During the second 1-week study period, 4-12 weeks later, participants will again ingest placebo solution (14 doses over 7 days). Blinding will occur by completely covering single-dose oral syringes with labels. 20% of participants will be randomized to this arm.
  Interventions: Drug: Placebo; Drug: Deuterated water (2H2O/D2O), 70%; Diagnostic Test: Insulin Suppression Test (IST)

INTERVENTIONS:
Drug: Placebo — Flavor-approximate placebo consisting of peppermint extract in diet tonic water, thickened with xanthan gum, provided in label-obscured single-use oral syringes at 40 µL per kg per dose. 80% of participants will receive placebo (14 doses over 7 days) during the first 1-week study period, while 20% of participants will receive an additional 14 doses of placebo over 7 days during the second study period, 4-12 weeks later.
  Other Names: Placebo solution
Drug: Diazoxide Oral Suspension, 2 mg per kg per dose — Eighty percent of participants will ingest diazoxide oral suspension at 2 mg per kg body weight per dose (14 doses over 7 days) during the study's second 1-week treatment period. Blinding will occur by completely covering single-dose oral syringes with labels.
  Other Names: Proglycem
  Arms: Placebo first, then Diazoxide
Drug: Deuterated water (2H2O/D2O), 70% — All participants will consume 18 aliquots of deuterated water (2H2O/D2O) 50 mL over 7 days during both study periods to assess hepatic de novo lipogenesis. Tracer enrichment will be determined in blood and saliva.
  Other Names: Heavy water
Diagnostic Test: Insulin Suppression Test (IST) — Participants receive intravenous infusions of regular insulin (32 milliunits [mU] per square meter [m2] per minute [min]), octreotide acetate (25 µg bolus + 0.27 µg/m2/min continuous infusion), and dextrose 20% in water (267 mg/m2/min continuous infusion) for 3 hours. Insulin resistance is reflected as the steady-state plasma glucose (SSPG) during the final 30 minutes of the procedure. IST is performed at the end of both study periods to determine the impact of placebo versus diazoxide on insulin sensitivity.

SUMMARY:
The goal of this clinical trial is to compare a one-week course of diazoxide (2 mg/kg per dose x 14 doses) and placebo in people with obesity and insulin resistance (IR) with metabolic dysfunction-associated steatotic liver disease (MASLD). The main question it aims to answer are how mitigation of compensatory hyperinsulinemia with diazoxide affects hepatic de novo lipogenesis, a major contributor to MASLD pathophysiology.

Participants will:

* Take 14 doses of placebo over 7 days, followed 4-12 weeks later by either 14 doses of diazoxide (at 2 mg per kg of body weight per dose [mpk]) or another 14 doses of placebo, over 7 days
* Take 18 doses of heavy (deuterated) water (50 mL each) over 7 days, twice
* Have blood drawn and saliva collected after an overnight fast on four mornings over the course of the study
* Undergo insulin suppression tests (IST) to assess the degree of insulin resistance at the end of each 1-week study period
* Consume their total calculated daily caloric needs as divided into three meals per day

Researchers will compare blood tests at the beginning and end of each 1-week study period in participants randomized (like the flip of a coin) to receive either placebo followed by diazoxide or placebo followed by placebo, to see how the drug treatment affects de novo lipogenesis, serum insulin, plasma glucose, and other serum lipid parameters (triglycerides, free fatty acids), among others.

DETAILED DESCRIPTION:
Metabolic dysfunction-associated steatotic liver disease (MASLD) is an under-appreciated complication of lipid dysmetabolism in type 2 diabetes (T2DM). Although it appears that insulin resistance (IR) is a mechanism common to both, the pathophysiology of its connection to unhealthy fat accumulation in the liver remains unclear. The investigators propose that the hyperinsulinemia that accompanies IR drives the excess hepatic de novo lipogenesis (DNL) that characterizes IR-associated MASLD. In other words, hepatic IR may be "selective," such that DNL is more sensitive to stimulation by insulin than is suppression of endogenous glucose production. As such, despite its potential impact on glucose metabolism, lowering insulin levels might attenuate the pro-steatotic drive in patients with IR. The investigators' objective, therefore, is to blunt endogenous insulin secretion using the insulin anti-secretagogue diazoxide in order to assess the impact on DNL.

This is a single-center, randomized, double-blinded, placebo-controlled, crossover clinical trial to determine the lipogenic impact of hyperinsulinemia reduction with diazoxide oral suspension in participants with obesity and insulin resistance (prediabetic state or elevated Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) score, + fasting hyperinsulinemia) who are diagnosed with MASLD. Participants will be randomized to one of two groups. Both groups will receive 14 doses of placebo over 7 days. Then, 4-12 weeks later, one group will cross over to receive 14 doses of diazoxide 2 mg per kg of body weight for 7 days, while the other group will receive a second 1-week course of placebo. Participants will consume heavy (deuterated) water for a total of 18 doses of 50 ml over each 1-week study period to measure de novo lipogenesis. They will present for outpatient blood draws and saliva collections after an overnight fast at the start and conclusion of each study period, and will undergo formal assessment of insulin resistance by the insulin suppression test (IST) at the end of each study period.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* Body mass index of 30-45 kg/m2
* Able to understand written and spoken English and/or Spanish
* Able to have pre-randomization screening labs drawn and study protocol initiated within 60 days of eligibility determination
* Presence of uncomplicated metabolic dysfunction-associated steatotic liver disease (MASLD) by vibration-controlled transient elastography (VCTE)

  * Steatosis score of S1-S3
  * Fibrosis score of F0-F2 (Note that if VCTE result is available from within past 6 months, then do not have to repeat VCTE for study purposes)
* Evidence of insulin resistance, represented by any or all of the following criteria:

  * Meeting either of the American Diabetes Association's definitions for prediabetes or impaired fasting glucose (IFG) on screening labs:

    * Prediabetes: Hemoglobin A1c 5.7-6.4%
    * IFG: plasma glucose of 100-125 mg dL-1 after ≥ 8-h fast
  * Homeostasis Model of Insulin Resistance (HOMA-IR) score ≥ 2.73
* Fasting hyperinsulinemia (fasting insulin level ≥ 13 μU/mL) on screening labs
* Written informed consent (in English or Spanish) and any locally required authorization (e.g., Health Insurance Portability and Accountability Act) obtained from the participant prior to performing any protocol-related procedures, including screening evaluations.

Exclusion Criteria:

* Unable to provide informed consent in English or Spanish
* Concerns arising at screening visit (any of the following):

  * Documented weight loss of ≥ 5.0% of baseline within the previous 3 months
  * Abnormal blood pressure (including on treatment, if prescribed)

    * Systolic blood pressure (SBP) < 90 mm Hg or > 160 mm Hg, and/or
    * Diastolic blood pressure (DBP) < 60 mm Hg or > 100 mm Hg
  * Resting heart rate < 55 bpm or ≥ 110 bpm
  * Abnormal screening electrocardiogram (or if on file, performed within previous 90 days)
  * Laboratory evidence of diabetes mellitus:

    * Hemoglobin A1c ≥ 6.5%, and/or
    * Fasting plasma glucose ≥ 126 mg/dL
  * Positive qualitative serum β-human chorionic gonadotropin (β-hCG, i.e., pregnancy test) in women of childbearing potential
  * Liver function abnormalities: transaminases (aspartate aminotransferase or alanine aminotransferase) > 3.0 x the upper limit of normal, and/or total bilirubin > 1.25 x the upper limit of normal
  * Abnormal screening fasting triglycerides > 500 mg/dL
  * Abnormal screening serum electrolytes that are considered clinically significant according to the clinical judgment of the PI
  * Creatinine equating to estimated glomerular filtration rate < 60 mL/min/1.73 m2
  * Abnormal screening blood counts (any of the following):

    * Hemoglobin < 10 g/dL
    * White blood cell count below the lower limit of normal for sex
    * Platelet count below the lower limit of normal for sex
  * Uric acid level above the upper limit of normal
* Reproductive concerns

  * Women currently pregnant (tested by serum and/or urine β-hCG)
  * Women currently breastfeeding
* Concerns related to glucose metabolism

  * History of having met any of the American Diabetes Association's definitions of diabetes mellitus (i.e., overt diabetes):

    * Hemoglobin A1c ≥ 6.5%
    * Plasma glucose ≥ 126 mg/dL after 8-h fast
    * Plasma glucose of ≥ 200 mg/dL at 2 h after ingestion of a 75-g glucose load
    * Random plasma glucose ≥ 200 mg/dL associated with typical hyperglycemic symptoms, diabetic ketoacidosis, or hyperglycemic-hyperosmolar state
  * History of gestational diabetes mellitus within the previous 5 years
  * Use of antidiabetic medications except metformin within the 90 days prior to screening
  * Clinical concern for absolute insulin deficiency (e.g., type 1 diabetes, pancreatic disease)
* Concerns related to lipid metabolism

  * Known diagnoses of familial hypercholesterolemia, familial combined hyperlipidemia, or familial hyperchylomicronemia
  * Use of fibrates, prescription-strength omega-3 fatty acids, or high-dose niacin within the 90 days prior to screening:
* Known, documented history (i.e., not to be newly screened/tested for study purposes), at the time of screening, of any of the following medical conditions:

  * Pancreatic pathology, including but not limited to neoplasia, pancreatitis, pancreatectomy
  * Cardiovascular disease (N.B. uncomplicated hypertension is not exclusionary)

    * Atherosclerotic cardiovascular disease: stable or unstable angina, myocardial infarction, ischaemic or hemorrhagic stroke, or transient ischaemic attack, peripheral arterial disease (claudication), use of dual antiplatelet therapy (aspirin + P2Y12 inhibitor), history of percutaneous coronary intervention
    * Heart rhythm abnormalities
    * Congestive heart failure of any New York Heart Association class
    * Symptomatic valvular heart disease (e.g., aortic stenosis)
    * Pulmonary hypertension
  * Chronic kidney disease, Stage 3 or higher (estimated glomerular filtration rate < 60 mL/min/ 1.73 m2), of any cause
  * Chronic liver disease other than uncomplicated MASLD, including but not limited to:

    * Advanced liver fibrosis, as determined by non-invasive testing, including fibrosis scores of F3-F4 on VCTE
    * Cirrhosis of any etiology
    * Autoimmune hepatitis or other rheumatologic disorder affecting the liver
    * Biliopathy (e.g., progressive sclerosing cholangitis, primary biliary cholangitis)
    * Chronic liver infection (e.g., viral hepatitis, parasitic infestation)
    * Hepatocellular carcinoma
    * Infiltrative disorders (e.g., sarcoidosis, hemochromatosis, Wilson disease)
  * Gout
  * Chronic infection with hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV)
  * Malabsorptive conditions
  * Active seizure disorder (including controlled with antiepileptic drugs)
  * Psychiatric diseases that are or have been decompensated within 1 year of screening, and/or require use of antipsychotic drugs associated with significant weight gain/metabolic dysfunction (e.g., clozapine, olanzapine), monoamine oxidase inhibitors, tricyclic antidepressants, or lithium
  * Known glucose-6-phosphate dehydrogenase (G6PD) deficiency
  * Other clinically significant endocrinopathies
  * Venous thromboembolic disease (deep vein thrombosis or pulmonary embolism) or any required use of therapeutic anticoagulation
  * Active malignancy, or hormonally active benign neoplasm, except allowances for non-melanoma skin cancer and differentiated thyroid cancer (Stage I only)
  * Clinical concern for increased risk of volume overload or hypotension (SBP <90 and/or DBP <60 mm Hg), including due to medications and/or heart/liver/kidney problems, as listed above
* Clinical concern for increased risk of volume overload or hypotension (SBP <90 and/or DBP <60 mm Hg), including due to medications and/or heart/liver/kidney problems, as listed above
* Use of certain medications currently or within 90 d prior to screening:

  * Prescribed medications used for any of the indications in the preceding list of excluded conditions, or their use within 90 d prior to screening, except allowances for:

    * Statins for primary prevention of cardiovascular disease
    * Use of drugs prescribed for indications other than the exclusionary diagnoses/purposes listed above (e.g., non-hydantoin antiepileptic drugs used for non-seizure indications, angiotensin converting enzyme inhibitor/angiotensin receptor blocker used for uncomplicated hypertension rather than for congestive heart failure, etc.)
    * Vasodilating drugs for any indication: hydralazine, nitrates, phosphodiesterase-5 inhibitors (e.g., sildenafil, tadalafil), minoxidil (oral)
    * Phenytoin or fosphenytoin for any indication
    * Oral or parenteral corticosteroids (at greater than prednisone 5 mg daily, or equivalent) for more than 3 days within the previous 90 days; topical and inhaled formulations are permitted
* History of certain weight-loss (bariatric) surgeries, including:

  * Roux-en-Y gastric bypass
  * Biliopancreatic diversion
  * Restrictive procedures (lap band, sleeve gastrectomy) performed within past year
* Clinical concern for alcohol overuse, including based on chart review and/or by participant's report of consuming more than 14 standard drinks per week for males or more than 7 standard drinks per week for females
* Regular use of tobacco, either daily or an average of at least 1 cigarette per day, and/or nicotine vaping more than 1 day per week
* Positive urine drug screen, except for lawfully prescribed medications or marijuana/tetrahydrocannabinol positivity, provided that the participant agrees not to use it during the same period that they will abstain from alcohol)
* Atypical circadian rhythm, such as due to night shift work, within 30 days of screening or expected within 30 days of each treatment period
* History of severe infection or ongoing febrile illness within 14 days of screening
* Any other disease or condition or laboratory value that, in the opinion of the investigator, would place the participant at an unacceptable risk and/or interfere with the analysis of study data.
* Known allergy/hypersensitivity to any component of the medicinal product formulations (including sulfa drugs), other biologics, intravenous (IV) infusion equipment, plastics, adhesive or silicone, history of infusion site reactions with IV administration of other medicines, or ongoing clinically important allergy/hypersensitivity as judged by the investigator.
* Concurrent enrollment in another clinical study of any investigational drug therapy or use of any biologicals within 5 half-lives of an investigational agent or biologic

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Hepatic de novo lipogenesis (absolute values) | Up to study day 7 during each 1-week study period
  Percent incorporation of newly synthesized fatty acids into serum or very low-density lipoprotein (VLDL) triglyceride (TG) (units: %)
Hepatic de novo lipogenesis (relative/change) | Up to study day 7 during each 1-week study period
  Percent incorporation of newly synthesized fatty acids into serum or VLDL TG (units: fold difference and/or ∆%)

SECONDARY OUTCOMES:
Fasting plasma/serum insulin (absolute values) | Up to study day 7 during each 1-week study period
  Measurement of fasting endogenous insulin levels during treatment with diazoxide 2 mpk vs. placebo (units: micro-international units [µIU] per mL).
Fasting plasma/serum insulin (relative/change) | Up to study day 7 during each 1-week study period
  Measurement of fasting endogenous insulin levels during treatment with diazoxide 2 mpk vs. placebo (units: fold difference and/or change in µIU/mL).
Fasting plasma glucose | Up to study day 7 during each 1-week study period
  Measurement of fasting plasma glucose levels during treatment with diazoxide 2 mpk vs. placebo (units: mg/dL).
Fasting serum or plasma triglycerides | Up to study day 7 during each 1-week study period
  Measurement of fasting plasma or serum triglyceride levels during treatment with diazoxide 2 mpk vs. placebo (units: mg/dL).
Fasting plasma free fatty acids | Up to study day 7 during each 1-week study period
  Measurement of fasting plasma free fatty acid levels during treatment with diazoxide 2 mpk vs. placebo (units: mmol/L).
Steady state plasma glucose (SSPG) during IST | At time points of 150, 160, 170, and 180 minutes during each 3-hour IST protocol
  Measurement of plasma glucose at 10-minute intervals during 30-minute steady-state period at the end of each IST (units: mg/dL)

OTHER OUTCOMES:
Skin de novo lipogenesis | Up to 3 hours during each IST
  Percent incorporation of newly synthesized fatty acids into sebum from healthy skin and, if present, skin from inflammatory skin lesions (units: %)
Deuterium tracer enrichment in body water (measured in blood) | Up to study day 7 during each 1-week study period
  Enrichment of total body water with deuterated water (2H2O/D2O) (units: %)
Deuterium tracer enrichment in body water (measured in saliva) | Up to study day 7 during each 1-week study period
  Enrichment of total body water with deuterated water (2H2O/D2O) (units: %)
Deuterium tracer enrichment in sebum | Up to 3 hours during each IST
  Enrichment of sebum with deuterated water (2H2O/D2O) (units: %)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua R Cook, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol